CLINICAL TRIAL: NCT06685978
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Phase III Clinical Trial of Efficacy and Safety of Xiangjurupining Capsule in the Treatment of Hyperplasia of Mammary Glands(Syndrome of Stagnation of Liver-qi and Phlegm)
Brief Title: Efficacy and Safety of Xiangjurupining Capsule for Hyperplasia of Mammary Glands
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-XJRPNJN-III
Record Dates: First submitted 2024-11-07; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Hyperplasia of Mammary Glands

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- :Xiangjurupining Capsule Placebo group (Placebo Comparator): Xiang Ju Ru Pi Ning capsule Placebo(0.45g per capsule ) 4 capsules each time,p.o.,tid,for 3menstrual cycle.
  Interventions: Drug: Xiang Ju Ru Pi Ning capsule Placebo
- Xiangjurupining Capsule Experimental group (Experimental): Xiang Ju Ru Pi Ning capsule (0.45g per capsule ) 4 capsules each time,p.o.,tid,for 3menstrual cycle.
  Interventions: Drug: Xiang Ju Ru Pi Ning capsule

INTERVENTIONS:
Drug: Xiang Ju Ru Pi Ning capsule Placebo — Xiang Ju Ru Pi Ning capsule Placebo(0.45g per capsule ) 4 capsules each time,p.o.,tid,for 3menstrual cycle.
  Other Names: Placebo group
  Arms: :Xiangjurupining Capsule Placebo group
Drug: Xiang Ju Ru Pi Ning capsule — Xiang Ju Ru Pi Ning capsule (0.45g per capsule ) 4 capsules each time,p.o.,tid,for 3menstrual cycle.
  Other Names: Experimental group
  Arms: Xiangjurupining Capsule Experimental group

SUMMARY:
This study will evaluate the efficacy and Safety of Xiangjurupining Capsule in the treatment of Hyperplasia of Mammary Glands(stagnation of liver-qi and phlegm).

DETAILED DESCRIPTION:
Xiangjurupiling Capsule is an oral pure Chinese medicine preparation.This study will evaluate the efficacy and Safety of Xiangjurupining Capsule in the treatment of Hyperplasia of Mammary Glands(stagnation of liver-qi and phlegm).

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18 to 50 (including boundary values);
2. Those who meet the diagnostic criteria for breast hyperplasia in Western medicine and have a disease course of more than 3 months;
3. Meets the traditional Chinese medicine differentiation criteria for liver depression and phlegm coagulation syndrome;
4. The BI-RADS grading of the target side breast ultrasound is 2-3 levels, while the BI-RADS grading of the non target side breast ultrasound is 1-3 levels;
5. During the screening period, the NRS score is ≥ 4 and there is a target mass detected by palpation;
6. During the introduction period, the average NRS score within the day of pain involvement is ≥ 4 points, and there is still the presence of the target mass on palpation;
7. During the import period, the number of days with pain involvement in the menstrual cycle is greater than 7 days;
8. With informed consent, voluntarily participate in the experiment and sign the informed consent form.

Exclusion Criteria:

1. Those who suffer from other breast diseases or breast pain caused by other reasons, such as mastitis, breast cancer, etc;
2. Patients with severe cardiovascular, cerebrovascular, liver, kidney, malignant tumors, hematological diseases, and psychiatric disorders;
3. Patients who have been previously diagnosed with dysfunctional uterine bleeding, amenorrhea, polycystic ovary syndrome, menopausal syndrome, hyperprolactinemia, Cushing's syndrome, and other diseases and still require treatment by adjusting hormone levels; Individuals who have been diagnosed with diseases that require long-term use of painkillers, such as dysmenorrhea, and are expected to be unable to stop using painkillers during the trial period.
4. Abnormal liver function (ALT or AST or ALP or GGT>1.2 times the upper limit of normal values) or abnormal kidney function (serum Cr or BUN or Urea>1.2 times the upper limit of normal values) that the researcher considers clinically significant and is not suitable for participation in clinical trials;
5. Women who are in pregnancy, lactation, menopause, or have a pregnancy plan within the past 6 months;
6. Chinese and western medicines and other therapies (including external application medicine, acupuncture and moxibustion, etc.) used to treat breast hyperplasia or relieve breast pain within 1 month or 5 half lives (whichever is the shortest) before screening and during the induction period, or contraceptives and sex hormone drugs have been used within half a year;
7. Individuals with severe menstrual cycle and/or menstrual irregularities (menstrual cycle>35 days or<21 days and/or menstrual period<3 days or>7 days);
8. Individuals with allergic constitution and known allergies to the components of the experimental drug prescription;
9. Suspect or have a history of alcohol and drug abuse;
10. Select patients who have participated in clinical trials and used investigational drugs within the previous month;
11. Failure to follow the physical contraceptive measures recognized by researchers for contraception;
12. According to the researchers' assessment, there may be other conditions or conditions that reduce the likelihood of inclusion or complicate the trial, such as frequent changes in the work environment that can lead to loss to follow-up, and individuals who cannot provide sufficient informed consent due to mental and behavioral disorders.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 430 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain relief rate | Baseline to the 3rd menstrual cycle
  Breast pain (NRS score) remission rate from baseline.Subject reported breast pain usingNRs( NumericalRatine Scalelscale onthe subiect daily diary.The NRS scale is a line composed of several points, marked with a scale of 0 to 10.The subjects rated themselves according to the most painful degree every day. The higher the score, the higher the degree of pain.

SECONDARY OUTCOMES:
Pain disappearance rate | Baseline to the 3rd menstrual cycle
  Breast pain (NRS score) disappearance rate from baseline.Subject reported breast pain usingNRs( NumericalRatine Scalelscale onthe subiect daily diary.The NRS scale is a line composed of several points, marked with a scale of 0 to 10.The subjects rated themselves according to the most painful degree every day. The higher the score, the higher the degree of pain.
Changes in mean NRS scores from baseline within days of pain involvement | Baseline to the 3rd menstrual cycle
  The mean value of breast pain per menstrual cycle was calculated from baseline.Subject reported breast pain usingNRs( NumericalRatine Scalelscale onthe subiect daily diary.The NRS scale is a line composed of several points, marked with a scale of 0 to 10.The subjects rated themselves according to the most painful degree every day. The higher the score, the higher the degree of pain.
Changes in maximum NRS scores from baseline | Baseline to the 3rd menstrual cycle
  Capture the highest value of breast pain per menstrual cycle from baseline.Subject reported breast pain usingNRs( NumericalRatine Scalelscale onthe subiect daily diary.The NRS scale is a line composed of several points, marked with a scale of 0 to 10.The subjects rated themselves according to the most painful degree every day. The higher the score, the higher the degree of pain.
Change in pain AUC (area under pain-time curve) from baseline | Baseline to the 3rd menstrual cycle
  The pain AUC was calculated from baseline based on the breast pain NRS score per menstrual cycle.
Change from baseline in days with NRS≥4 points | Baseline to the 3rd menstrual cycle
  The number of days in each menstrual cycle with an NRS score greater than 4 for breast pain was captured from baseline.Subject reported breast pain usingNRs( NumericalRatine Scalelscale onthe subiect daily diary.The NRS scale is a line composed of several points, marked with a scale of 0 to 10.The subjects rated themselves according to the most painful degree every day. The higher the score, the higher the degree of pain.
Within a few days of pain involvement within a menstrual cycle, the average NRS score decreased by 70% from baseline. | Baseline to the 3rd menstrual cycle
  The mean NRS score decrease from baseline within days of pain involvement was 70%.Subject reported breast pain usingNRs( NumericalRatine Scalelscale onthe subiect daily diary.The NRS scale is a line composed of several points, marked with a scale of 0 to 10.The subjects rated themselves according to the most painful degree every day. The higher the score, the higher the degree of pain.
TCM syndrome scores | the 3rd menstrual cycle after treatment
  Compared wth baseline;the scores of changes ofTCM syndrome Evaluaion at each visit .This instrument consists oftwo primary symptoms:breast pain,breast mas ,and foursecondary symptoms.fourlevels to measure severtyof primarysymptoms (0.2、4、6) and secondarysymptoms (0、1、2.3),respectively. Record the tongue and pulseconditions. The TCM syndrome efect calculated bynimodipine method. The final score has a rangeof0 to 100. The efect ofTCM syndrome from 0% negative) to 100%(disappear).
SF-36V2 | the 3rd menstrual cycle after treatment
  Changes in SF-36 V2 scale scores and total scores from baseline.The SF-36 scale is a universal scale developed by the American medical research group to assess the quality of life (17 Appendix: SF-36 v2 rating scale), which is widely recognized and used in the world. The SF-36 v2 scale includes 36 entries that assess health-related quality of life in eight dimensions: physiological function (PF), physiological function (RP), physical pain (BP), general health (GH), vitality (VT), social function (SF), emotional function (RE), and mental health (MH). A Health Change (HT) entry is also included. The quality of life was retrospectively evaluated by the participants at visit 2, visit 5 and visit 6. The higher the score, the higher the quality of life. The results of V2 examination were used as the baseline to calculate the scores of all dimensions of quality of life and the total score.
The target lump | the 3rd menstrual cycle after treatment
  Assess the scope the size and the hardness of the tareet lump by palpation.The doctor palpated the breast ofthe subjects and measured the size of the target lump with a ruler .Four quadrant method was used to record the number of the target lump's quadrants. Four level(0.2.4.6)to measure The scope,the size and the hardness of lump .The score from 0(none) to 6(most severe).
The target lump area | the 3rd menstrual cycle after treatment
  Assess the breast glandular section thickness and nodules of the target lump area by B-ultrasound.

CONTACTS AND LOCATIONS:
Locations (27):
- China (27):
  - Dongzhimen Hospital, Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - East Hospital of Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Guang 'anmen Hospital, Beijing, Beijing Municipality
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing, Chongqing Municipality
  - Xiamen Hospital of Traditional Chinese Medicine, Xiamen, Fujian
  - Guangdong Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Guang 'anmen Hospital Baoding Hospital, Baoding, Hebei
  - Cangzhou Hospital of Integrated Chinese and Western Medicine, Cangzhou, Hebei
  - Hebei Provincial Hospital of Traditional Chinese Medicine, Shijiazhuang, Hebei
  - Oilfields General Hospital in Daqing, Daqing, Heilongjiang
  - Luoyang Third People's Hospital, Luoyang, Henan
  - Zhengzhou People's Hospital, Zhengzhou, Henan
  - Wuhan Third Hospital, Wuhan, Hubei
  - The First Affiliated Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - The First Affiliated Hospital of Hunan College of Traditional Chinese Medicine (Hunan Provincial Direct Hospital of Traditional Chinese Medicine), Zhuzhou, Hunan
  - Jiangsu Provincial Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - North Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - The Second Affiliated Hospital of Shandong First Medical University, Taian, Shandong
  - Weifang Hospital of Traditional Chinese Medicine, Weifang, Shandong
  - Longhua Hospital affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shanxi Hospital of Traditional Chinese Medicine, Taiyuan, Shanxi
  - The First Affiliated Hospital of Tianjin University of Chinese Medicine, Tianjin, Tianjin Municipality
  - Urumqi maternal and child Health Care Hospital, Ürümqi, Xinjiang
  - Zhejiang Provincal Hospital of TCM, Hangzhou, Zhejiangsheng

IPD SHARING:
Plan to Share IPD: No